CLINICAL TRIAL: NCT03464396
Title: Physiologic Biomarkers Predicting Ventilatory Instability and Hypoxemia in Pre Mature Infants
Brief Title: Prematurity-Related Ventilatory Control
Acronym: PreVent
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201611138; 5U01HL133700-02 (NIH)
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Respiratory Control in Premature Infants
Keywords: Periodic breathing; Apnea of prematurity; Chronic Lung disease; Prematurity; Respiratory disease; Hypoxia; Pulmonary Hypertension
MeSH Terms: conditions — Apnea; Premature Birth; Respiration Disorders; Hypoxia; Hypertension, Pulmonary | interventions — Magnetic Resonance Imaging; Echocardiography; Caves; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal Swabs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infant study visits: Preterm infants Study Visits
  1. Bedside Physiology Study at 28, 32, 36, 40, and 52 weeks GA.
  2. Respiratory tests:
     * Carotid Body Function Test will be completed at 32, 36, 40 and 52 weeks GA
     * Room Air Challenge (RAC) or Hypoxia Challenge Test (HCT) will be completed at 36 weeks GA
     * Effects of nasal cannula flow be completed at 28, 32, 36, 40 and 52 weeks GA
  3. Magnetic Resonance Imaging (MRI): Completed on a subset of infants between 37-40 weeks GA or before discharge, whichever comes first.
  4. Echocardiogram (Echo): Completed at 32, 36 and 52 weeks GA
  5. Blood sample: Obtained at 32, 36 and 52 weeks GA
  Interventions: Other: Bedside Physiology study; Other: Carotid Body Function Test; Other: Room Air Challenge; Other: Hypoxia Challenge Test; Other: Effects of Nasal Cannula Flow; Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Echocardiogram; Other: Blood Sample

INTERVENTIONS:
Other: Bedside Physiology study — A 90-minute recording in conjunction with the respiratory evaluations using standard recording equipment that includes a conventional pulse oximeter, an EEG, an airflow sampling catheter near the nose, and respiratory inductance plethysmography (RIP) bands. Standard clinical bedside monitoring will continue during the respiratory evaluations.
Other: Carotid Body Function Test — Infants without nasal cannula will have a nasal cannula placed in their nares. After a 15-minute baseline period and during quiet sleep, the infant will then be exposed to 30 seconds of 100% oxygen (O2) by increasing FiO2. This test will be repeated 3 times, with at least 3 minutes between tests to allow for return of oxygen saturation (SpO2) to baseline values. If oxygen saturations increase to 99% for 15 seconds or the infant is apneic for greater than 5 seconds following initiation of 100% oxygen (O2), the test will be stopped and FiO2 brought back to baseline. Infants in the NICU will be monitored continuously with heart rate, respiratory rate, and SpO2% for 12 hours after Carotid Body Function Test according to NICU standards. Infants discharge who return for Carotid Body Function Test at 40 and 52 weeks PMA will be monitored continuously for 1 hour after the test is finished.
Other: Room Air Challenge — Infants receiving nasal cannula high flow support 3 liters per minute (LPM) or less with or without supplemental O2 at 36 weeks PMA will be eligible. After a 15-minute quiet sleep period, infants' FiO2 will be weaned, in 0.20 decrements for 5 min intervals. Flow then decreased in 10 min intervals, initially in 1 Liter Per Minute (LPM) decrement until nasal cannula flow is 1LPM, and then decreased by 50% decrements to 0.125 LPM then off. If the infant is weaned to room air alone for 15 minutes, not meeting failure criteria, he/she has passed the RAC. Failure of the RAC is defined as occurring when SpO2% falls below 80%, even briefly, or remains less than 90% for 5 consecutive minutes any time during the test, bradycardia (Heart rate [HR] < 80 bpmx 10 sec) or persistent apnea despite stimulation. Infant is returned to the level of support provided before the RAC begun if meets any failure criteria.
  Other Names: RAC
Other: Hypoxia Challenge Test — A physician investigator will review 30 minutes of continuous recording made 24 hours prior to test scheduled to identify infants that are at high risk for significant oxygen desaturations during Hypoxemia Challenge.
  If subject passes the screening test, the hypoxic challenge will be performed. For the hypoxemia test, a nasal cannula will be placed prior to a 15 minute period of quiet sleep recorded to confirm antecedent stability of ventilatory pattern and SpO2%. During the 15 minutes of quiet sleep, the infant is required to maintain a SpO2 of > 92% in order to undergo the HCT. After the 15-minute baseline recording, HCT will begin using FiO2 = 0.18 for 5 minutes, unless failure criteria is met: SpO2% < 80% even briefly, or SpO2% 80% to 85% for 15 seconds. If infant does not meet failure criteria, infant will be given FiO2 0.15 for 10 minutes. If an infant meets even a single criterion for failure, Hypoxic mixture will be stopped.
  Other Names: HCT
Other: Effects of Nasal Cannula Flow — Infants will have nasal catheter in place (NeoTech Premature RAM Cannula). A 15-minute baseline recording of physiologic study parameters prior to initiation. Tested in three groups of infants.
  1. 28 and 32 weeks PMA flow rates increased after a 15-minute baseline period to 3LPM, or by 1LPM to a max of 5LPM for 15 minutes. Infant on Bubble CPAP will be increased 1cm H2O to max 8 cm H2O for 15 minutes.
  2. Infant's that fail the RAC or HCT at 36 weeks with periodic breathing, high flow at 3LPM will be started for 2 minutes or until periodic breathing stops. Infants on Bubble CPAP will not undergo the RAC or HCT. Their pressure is increased by 1cm H20 to max of 8 cm H2O for 15 minutes.
  3. Infant on RA at 40 and 52 weeks PMA with periodic breathing lasting longer than 1 minute during the 15-minute baseline period, flow at 3LPM will be started for 2 minutes or until periodic breathing stops.
Diagnostic Test: Magnetic Resonance Imaging — A non-sedating MRI scan will be performed on 3 subsets of infants at 37-40 weeks Post Menstrual Age (PMA), or when infant is within one week of discharge from the NICU. Standard images as well as research images will be obtained. The research images use the same MRI scanner and collection techniques as standard clinical imaging, but provide a more detailed examination of brain anatomy and injury. Collection of these sequences using our standard non-sedated acquisition practices for infants is well tolerated. Infants will be placed in scanner by registered nurse accompanied by radiology technician to assure infants' comfort during scan. Infant will remain on cardio-respiratory monitor during MRI via a pulse oximetry probe. It will take no longer than one hour to complete MRI scan including transportation to radiology unit.
  Other Names: MRI
Diagnostic Test: Echocardiogram — An echocardiogram (referred to as an ultrasound of the heart on the consent form) will be performed to assess cardiac structure and function. Echocardiograms are performed routinely in premature newborns in the NICU. The Echocardiogram will be performed at the infant bedside and will be coordinated with bedside nurse. The infant will remain on a cardio-respiratory monitor during the echocardiogram for approximately 15 minutes.
  Other Names: Echo
Other: Blood Sample — Infants that have echocardiograms will have a blood sample collected near the time the echocardiogram is obtained, 3-blood samples total. The blood sample will only be collected with parental permission on an opt-in or out-basis and collected only with routine clinical labs.

SUMMARY:
The purpose of this research study is to improve our understanding of unstable breathing and heart blood flow patterns seen in premature infants. The investigator will use novel non-invasive measures to understand the determinants of these unstable breathing and heart flow patterns to potentially identify new therapies for their prevention.

DETAILED DESCRIPTION:
The investigator will look at results of breathing tests, non-invasive sound wave (ultrasound) test of the heart and blood vessel (Echocardiography), and a sample of blood to see if it is possible for early detection of breathing control and lung blood vessel dysfunction (pulmonary vascular disease) in infants that are at risk for exposure to long term low oxygen levels. A subset of infants will have a magnetic resonance Imaging study (MRI) between 37- 40 weeks gestational age (GA) or at the time of discharge, whichever comes first.

Respiratory tests include:

* Bedside Physiology Study completed at 28, 32, 36, 40, and 52 weeks GA in conjunction with the respiratory tests. A 90-minute recording will be made using standard recording equipment that includes a conventional pulse oximeter, an EEG, an airflow sampling catheter near the nose, and respiratory inductance plethysmography (RIP) bands. Standard bedside monitoring will continue during the physiologic studies
* Carotid Body Function Test completed at 32, 36, 40 and 52 weeks GA. This test is to unmask respiratory instability in response to hyperoxia.
* Challenge Test completed at 36 weeks GA.

  1. Infants receiving nasal cannula flow with or without supplemental oxygen will undergo a Room Air Challenge Test.
  2. Infants on RA alone will undergo a Hypoxia Challenge test.
* Effects of Nasal Cannula Flow completed at 28, 32, 36, 40 and 52 week's GA. The flow will be increased through a nasal cannula. This test is to see how flow effects the breathing pattern.

A subset of infants will have an MRI between 37-40 weeks GA or before discharge, whichever comes first. The MRI will allow the doctors to look and see if there is any injury present in the brain that can be linked to an abnormal breathing pattern called periodic breathing.

A subset of infants will have an Echocardiogram (Echo) at 32, 36 and 52 weeks GA. The Echo is performed to assess cardiac structure and function. Echocardiography is performed routinely in premature newborns in the Neonatal Intensive Care Unit (NICU). The echocardiogram will be performed at the infant bedside and will be coordinated with bedside nurse. The infant will remain on a cardio-respiratory monitor during the echocardiogram for approximately 15 minutes.

Infants that have an Echo will have a blood sample collected near the time of the Echo, 3-blood samples total. The purpose of collecting the blood sample is to detect if the Fibroblast Growth Factor (FGF2) level is elevated and possibly be a biomarker of early pulmonary hypertension in pre term infants validated with the echo.

ELIGIBILITY:
Inclusion Criteria:

* All infants born between 24 0/7 and 28 6/7 weeks GA admitted to the Neonatal Intensive Care Unit at St. Louis Children's Hospital will be considered for enrollment.

Exclusion Criteria:

* Infants not likely to survive
* Infant with significant heart disease
* Infant with a significant congenital abnormalities of the central nervous system, nose, mouth lungs or ribs, or congenital diseases that affect lung growth
* Physician refusal
* Unlikely that the infant will be available for 52-week follow-up visit.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants admitted to the Neonatal Intensive Care Unit who are born between 24 0/7 to 28 7/8 weeks GA
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Respiratory phenotype based on physiologic testing | 36 weeks post menstrual age
  Categorization of subjects based on physiologic Challenge Tests into one of four respiratory phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: James Kemp, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coste F, Ferkol T, Hamvas A, Cleveland C, Linneman L, Hoffman J, Kemp J. Ventilatory control and supplemental oxygen in premature infants with apparent chronic lung disease. Arch Dis Child Fetal Neonatal Ed. 2015 May;100(3):F233-7. doi: 10.1136/archdischild-2014-307272. Epub 2015 Feb 25. PMID 25716677
- [Background] Carroll JL, Agarwal A. Development of ventilatory control in infants. Paediatr Respir Rev. 2010 Dec;11(4):199-207. doi: 10.1016/j.prrv.2010.06.002. Epub 2010 Jul 31. PMID 21109177
- [Derived] Mammel DM, Carroll JL, Warner BB, Edwards BA, Mann DL, Wallendorf MJ, Hoffmann JA, Conklin CM, Pyles H, Kemp JS. Quantitative and Qualitative Changes in Peripheral Chemoreceptor Activity in Preterm Infants. Am J Respir Crit Care Med. 2023 Mar 1;207(5):594-601. doi: 10.1164/rccm.202206-1033OC. PMID 36173816